CLINICAL TRIAL: NCT06040229
Title: Mechanism of Children With Relapsed and Refractory Rhabdomyosarcoma (RMS)
Brief Title: Retrospective Study in FFPE Samples From Younger Patients With Rhabdomyosarcoma
Status: Completed | Type: Observational
Sponsor: Shandong First Medical University (Other)
Collaborators: Shandong Tumor Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: Children's Oncology Group
Record Dates: First submitted 2023-09-10; First posted 2023-09-15 (Actual); Last update posted 2023-09-15 (Actual); Status verified 2023-09

CONDITIONS: Alveolar Childhood Rhabdomyosarcoma; Embryonal Childhood Rhabdomyosarcoma; Recurrent Childhood Rhabdomyosarcoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — FFPE samples
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This retrospective study is looking into mechanisms of drug therapy resistance in FFPE samples in recurrent and refractory Rhabdomyosarcoma (RMS) in pediatric patients who have experienced lung recurrence. The study employs advanced techniques such as single-cell transcriptomics and spatial transcriptomics to gain a comprehensive understanding of these mechanisms.

DETAILED DESCRIPTION:
This research seeks to enhance our understanding of drug resistance mechanisms in recurrent and refractory RMS in pediatric patients, particularly in the context of lung recurrence. The utilization of cutting-edge techniques like single-cell transcriptomics and spatial transcriptomics allows for a more in-depth and comprehensive analysis of the molecular and spatial aspects of drug resistance in this challenging pediatric cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Pediatric Patients: Participants in this study should be pediatric patients, typically defined as individuals aged from infancy to 18 years old, who have been diagnosed with recurrent and refractory Rhabdomyosarcoma (RMS).
2. Lung Recurrence: Included patients must have a documented history of lung recurrence of RMS as a specific clinical manifestation.
3. Availability of FFPE Samples: Patients for whom formalin-fixed paraffin-embedded (FFPE) tissue samples are available for analysis are eligible for inclusion.

Exclusion Criteria:

1. Other Histological Types: Patients with RMS of histological subtypes other than those relevant to the study focus are excluded.
2. Incomplete Clinical Data: Patients with incomplete or insufficient clinical data necessary for the study's objectives may be excluded to ensure robust analysis and interpretation of results.

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: All participants have previously been diagnosed with RMS, a rare and aggressive form of pediatric soft tissue cancer. Importantly, their RMS cases are characterized by recurrence, indicating that the cancer has returned after initial treatment, and refractoriness, meaning it has not responded well to standard therapies.
  A defining feature of the study population is the presence of documented lung recurrence. This signifies that the RMS has re-emerged specifically within the lung tissue. Lung recurrence is a critical clinical aspect being investigated in this study.
Sampling Method: Non-Probability Sample
Enrollment: 6 (Actual)
Dates: Start 2023-04-01 (Actual); Primary Completion 2023-07-01 (Actual); Study Completion 2023-09-01 (Actual)

PRIMARY OUTCOMES:
Gene expression pattern | 2023.12.31
  Identification and characterization of specific genetic alterations and gene expression patterns associated with drug therapy resistance in recurrent and refractory Rhabdomyosarcoma (RMS) in pediatric patients, particularly in cases of lung recurrence, using single-cell transcriptomics and spatial transcriptomics.

CONTACTS AND LOCATIONS:
Overall Officials: Tao Xu, Principal Investigator — Shandong First Medical University
Locations (1):
- Jinan central hospital affiliated to Shandong First Medical University, Jinan, Shandong, China

IPD SHARING:
Plan to Share IPD: Undecided